CLINICAL TRIAL: NCT07060612
Title: Incidencia y Factores de Riesgo Para el Desarrollo de infección fúngica Invasiva en Pacientes Con diagnóstico de Leucemia mieloblástica Aguda
Brief Title: Incidence and Risk Factors for the Development of Invasive Fungal Infection in Patients Diagnosed With Acute Myeloblastic Leukemia (HIFA)
Acronym: HIFA
Status: Active, not recruiting | Type: Observational
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0322-1
Record Dates: First submitted 2025-06-09; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: AML
Keywords: Fungal; AML

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients diagnosed with acute myeloblastic leukemia (AML) who receive intensive chemotherapy treatment have a high incidence of invasive fungal infection (IFI). IFI is a significant cause of morbidity and mortality in this population. Its diagnosis is generally challenging, leading to delays in treatment initiation and a worse prognosis. Various strategies have been proposed to improve outcomes: prophylaxis, empirical treatment, and preemptive strategies, but the optimal approach remains unknown.

Several authors advocate for tailoring IFI control strategies based on local IFI incidence and the risk factors present in each epidemiological area. In AML patients treated at our center, a thorough understanding of IFI incidence, associated risk factors, and the strategies adopted for its control during different historical periods will allow us to optimize patient management in the future to improve outcomes.

To this end, the investigators propose conducting a retrospective epidemiological study that captures routine clinical practice in the management of IFI at our center from January 1, 2015, to December 31, 2024. This study will record data on diagnosis, patient characteristics, and the development of IFI, regardless of age or treatment received.

Secondarily, the investigators aim to determine the incidence and epidemiological characteristics of IFI in this population, identify and confirm risk factors, and retrospectively evaluate the diagnostic and control strategies adopted for IFI across different historical periods. The study design will be retrospective, documenting routine IFI management practices at our center. No diagnostic or therapeutic interventions will be performed. All patients diagnosed with AML from January 1, 2015, to December 31, 2024, will be included, regardless of AML subtype, disease progression, or treatment received. Data will be collected on key AML characteristics at diagnosis, treatment received and number of cycles, IFI diagnosis according to the 2008 EORTC/MSG criteria, and the management of this complication.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with AML regardless of the treatment received (first line and relapsed/refractory).

Patients older than 15 years (adult unit) No contraindications for antifungal therapy/prophylaxis.

Exclusion Criteria:

* Patients with acute promyelocytic leukemia (APL). Patients with insufficient data (not evaluable).

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive unselected patients with AML diagnosed at the Hospital Universitario y Politécnico La Fe between 2015 and 2024. Clinical records of all patients will be reviewed to assess their eligibility for this retrospective study
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Primary objectives | 9 years
  To evaluate the incidence and risk factors for the development of IFI/BIFD in patients diagnosed with AML, regardless of the treatment received (first-line and relapsed/refractory patients).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario y Politécnico La Fe, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided